CLINICAL TRIAL: NCT00991549
Title: Comparative Evaluation of the Effectiveness of 2 Available Resources in Estrie, for the Prevention of Type 2 Diabetes in High-risk Subjects
Brief Title: Diabetes Prevention In Estrie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other); Novonordisk endocrine fellowship program (Unknown)
Responsible Party: Dr Marie-France Langlois, Universitaire de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04-087
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Overweight; Glucose Intolerance
Keywords: overweight; obesity; glucose intolerance; pre-diabetes
MeSH Terms: conditions — Overweight; Glucose Intolerance; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): interdisciplinary weight loss intervention
  Interventions: Behavioral: interdisciplinary intervention or meeting-seminars
- 2 (Active Comparator): Small group seminars without interdisciplinary intervention
  Interventions: Behavioral: interdisciplinary intervention or meeting-seminars

INTERVENTIONS:
Behavioral: interdisciplinary intervention or meeting-seminars — one-year individualized interdisciplinary weight loss program vs. small group seminars on healthy lifestyle

SUMMARY:
This study compared the efficacy at one year of an interdisciplinary approach including individual counseling and group seminars versus group seminars alone to induce weight loss in subjects at high risk of developing type 2 diabetes.

This study also compare if a participant's presence in small informative meeting groups as the only form of intervention is sufficient to induce a lifestyle change, thus inducing the weight loss needed for the prevention of the diseases associated with obesity.

DETAILED DESCRIPTION:
Eligible participants will be randomized into 2 intervention groups (30 per group):

1. Small Meeting groups: a curriculum of 25 meeting-seminars will take place for 45 minutes, each one approaching various aspects of nutrition, physical activity, psychology, motivation and medical needs. These seminars are administered by the professionals of the obesity clinic and are already in place. However, these are usually only offered to the patients registered with the obesity clinic.
2. Obesity Clinic of CHUS: combination of 25 described meeting-seminars see-high, in addition to individual interviews every 6 weeks with the interdisciplinary team of the obesity clinic of CHUS (usual operation).

Subjects will be evaluated initially and then every 3 months during 1 year by the following measurements: questionnaires to evaluate motivation and physical activity; 3 day dietary journals; weight assessment, using both metabolic and mechanical balance; waist circumference; and blood pressure.

A medical evaluation with size measure, a test evaluating knowledge of the participants on obesity, OGTT (Oral Glucose Tolerance Test) - a 5 hour determination of secretion and resistance to insulin, insulin-mediated suppression of plasma non-esterified fatty acids, a plasma lipid profile, accelerometry, bio electric impedance, and an activity physical test (6 minute walk test) will be carried out initially, and then repeated for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* pre diabetic state underlined by a marginal fasting glycemia between 6,1 and 6,9 mmol/L and/or a glucose intolerance with glucose confirmed by an OGTT 2 hours
* overweight or obesity (BMI > 27 kg/m² ; (Body Mass Index))
* enlightened assent

Exclusion Criteria:

* Impossibility to be present at the visits
* Physical/motor incapacity (or other) making one unable and/or insecure to walk at a moderate to rapid speed of 6 min and more
* Use of an anti-obesity treatment during the last 3 months
* Bariatric Surgery in the past
* Planned Pregnancy
* Pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-12; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
a weight loss of 7% in at least 19% of the subjects | one year
reduced body weight of at least 5.6 kg in at least 25% of the subjects | one year
an increase in the level of physical activity by at least 150 minutes per week in at least 29% of the subjects | one year
a reduced daily caloric intake of at least 450 kcal/jour in at least 25% of the subjects | one year
a reduced percentage of the calories introduced in the form of fat of at least 6.6%, in absolute value, in at least 25% of the subjects | one year

SECONDARY OUTCOMES:
change in insulin sensitivity by HOMA | one year
change in insulin secretion during an OGTT by deconvolution of plasma c-peptide | one year
change in beta cell function by calculation of the disposition index | one year
change in insulin-mediated suppression of plasma non-esterified fatty acids during an OGTT | one year
relation between weight loss and change in insulin sensitivity, beta cell function, and insulin-mediated suppression of plasma non-esterified fatty acids | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Medecine department, Division of endocrinology, CHUS
Locations (1):
- Centre de Recherche Clinique (CRC), Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Gagnon C, Brown C, Couture C, Kamga-Ngande CN, Hivert MF, Baillargeon JP, Carpentier AC, Langlois MF. A cost-effective moderate-intensity interdisciplinary weight-management programme for individuals with prediabetes. Diabetes Metab. 2011 Nov;37(5):410-8. doi: 10.1016/j.diabet.2011.01.003. Epub 2011 Apr 13. PMID 21489843